CLINICAL TRIAL: NCT01581034
Title: A Randomized, Placebo-controlled, Double-blinded Trial on the Effect of PADMA 28 on Endothelial Function, Biomarkers and the Autonomic Nervous System in Patients With Coronary Artery Disease
Brief Title: Effect of PADMA 28 on Endothelial Function, Autonomic Nervous System and Biomarkers in Patients With Coronary Artery Disease
Acronym: PADMA 28
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: 146/11
Record Dates: First submitted 2012-04-16; First posted 2012-04-19 (Estimated); Last update posted 2013-08-01 (Estimated); Status verified 2013-07

CONDITIONS: Coronary Artery Disease
Keywords: endothelial function; biomarkers; autonomic nervous system; coronary artery disease
MeSH Terms: conditions — Coronary Artery Disease | interventions — Padma 28

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Padma (Active Comparator)
  Interventions: Drug: PADMA 28
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: PADMA 28 — PADMA 28 is a biological drug registered in Switzerland. It contains 20 herbs from Tibet. 3 times 2 capsules per day (30min to 1h before breakfast, lunch and dinner) of PADMA 28 or placebo will be taken. One capsule contains 403mg.
  Arms: Padma
Drug: Placebo — 3 times 2 capsules per day (30min to 1h before breakfast, lunch and dinner) of placebo will be taken. One capsule contains 403mg.
  Arms: Placebo

SUMMARY:
This randomized, placebo-controlled, double-blinded trial investigates the effect of a 6 week intake of PADMA 28 on the endothelial function, biomarkers and the autonomic nervous systems in patients with coronary artery disease. The investigators hypothesize that PADMA 28 has a beneficial effect on endothelial function, arterial stiffness, the autonomic nervous systen and the blood inflammatory markers in patients with coronary artery disease compared to placebo treatment.

DETAILED DESCRIPTION:
Background

This randomized, placebo-controlled, double-blinded trial investigates the effect of a 6 week intake of PADMA 28 on the endothelial function, biomarkers and the autonomic nervous systems in patients with coronary artery disease. PADMA 28 contains 20 herbs from Tibet. The endothelial function will be measured by EndoPAT 2000, the autonomic nervous system by an ambulatory electrocardiography during the orthostatic reaction and the biomarkers will be analyzed with taking a blood sample. The investigators hypothesize that PADMA 28 has a beneficial effect on endothelial function, arterial stiffness, the autonomic nervous systen and the blood inflammatory markers in patients with coronary artery disease compared to placebo treatment.

Objective

To assess the effect of PADMA 28 on endothelial function, autonomic nervous system and biomarkers in patients with coronary artery disease.

Methods

80 patients with coronary artery disease will be recruited for the study. To measure endothelial function, the investigators use EndoPAT 2000. The autonomic nervous system will be analysed with ambulatory electrocardiography.

ELIGIBILITY:
Inclusion Criteria:

* Male patient with coronary artery disease
* Stable medication
* Physically stable
* Psychologically stable
* Written informed consent
* Willing and able to comply with all trial requirements
* Must have completed rehabilitation program since at least 6 months and no longer than 5 years prior to study begin

Exclusion Criteria:

* Acute coronary syndrome within the last three months
* Abnormal high hepatic enzymes
* Renal insufficiency with compensated retention
* Intake of medication which may affect endothelial function
* Currently smoking
* Current malignant diseases, which may reduce the expectancy of life
* Chronic heart failure
* Insulin-dependent diabetes
* Known hypersensitivity against any ingredient of PADMA 28
* Longterm intake of supplements
* Serious mental health issues
* Alcohol and/or drug abuse
* Simultaneous participation in another clinical trial

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2012-04; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Endothelial function | At completion of the study, expected to be at 6 weeks
  Expressed as Reactive Hyperemic Index (RHI), measured by non-invasive peripheral arterial tonometry

SECONDARY OUTCOMES:
Autonomic nervous system | At completion of the study, expected to be at 6 weeks
  Cardiac autonomic tone (expressed as frequency domain parameters of heart rate variability (HRV) & measured by ECG)
Biomarkers in blood | At completion of the study, expected to be at 6 weeks
  Blood inflammatory and anticoagulative biomarkers, measured by fasting blood samples

CONTACTS AND LOCATIONS:
Overall Officials: Hugo Saner, Prof. Dr., Study Chair — Department of cardiovascular prevention and rehabilitation, Bern University Hospital
Locations (1):
- Swiss Cardiovascular Prevention and Rehabilitation Center, Bern University Hospital, Bern, Switzerland

REFERENCES:
- [Derived] Schafer D, Lambrecht J, Radtke T, Wilhelm M, Saner H. Effect of a Tibetan herbal mixture on microvascular endothelial function, heart rate variability and biomarkers of inflammation, clotting and coagulation. Eur J Prev Cardiol. 2015 Aug;22(8):1043-5. doi: 10.1177/2047487314544985. Epub 2014 Sep 10. PMID 25208904